CLINICAL TRIAL: NCT03695653
Title: Tailored Adaptive Mobile Messaging to Reduce Problem Drinking
Brief Title: Messaging Interventions to Reduce Alcohol Problems Project
Acronym: MIRAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Partnership to End Addiction (Other)
Collaborators: Feinstein Institute for Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01AA025058 (NIH)
Record Dates: First submitted 2018-09-28; First posted 2018-10-04 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2020-07

CONDITIONS: Alcohol-Related Disorders; Alcohol Use Disorders; Alcohol Drinking; Alcoholism; Alcohol Abuse
Keywords: Drinking; Alcohol Problems; Moderation-Oriented Treatment; Controlled Drinking; Reduced Drinking; Problem Drinking; Text Message; Mobile Phone; Technology
MeSH Terms: conditions — Alcohol-Related Disorders; Alcoholism; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drink Tracking (MA) Condition (Active Comparator): Ps will receive weekly mobile assessment trick tracking described above for six months in addition to the guidelines on safe drinking.
  Interventions: Behavioral: Drink Tracking (MA)
- TA Intervention (Experimental): The TA intervention is tailored but will adapt over time too
  Interventions: Behavioral: Adaptive Tailored (TA)
- Tailored Content Only (TO) (Experimental): The TO treatment arm includes tailored text messages sent at 6pm daily based on the baseline assessment.
  Interventions: Behavioral: Tailored (TO)

INTERVENTIONS:
Behavioral: Drink Tracking (MA) — Weekly drink tracking for self-monitoring and assessment
  Arms: Drink Tracking (MA) Condition
Behavioral: Adaptive Tailored (TA) — Messages are sent more frequently and tailored to some baseline characteristics and adapt to progress
  Arms: TA Intervention
Behavioral: Tailored (TO) — Messages are sent more frequently and tailored to some baseline characteristics
  Arms: Tailored Content Only (TO)

SUMMARY:
The study is designed to develop and test a tailored adaptive text messaging/short message service (SMS) intervention for individuals interested in reducing their alcohol consumption.

According to the National Institute on Alcohol Abuse and Alcoholism, problem or risky drinking is defined as greater than 7 standard drinks per week for women and 14 standard drinks per week for men. Other groups have other criteria (e.g., 10 drinks for women and 14 for men per week). The Institute of Medicine reports that problem drinkers are those with mild-to-moderate problem severity who do not have physical dependence.

Heavy drinking individuals with non-abstinence goals rarely seek treatment for excessive alcohol use, and newer methods such as internet screening and mobile apps provide opportunities to engage and treat this difficult to reach population. There are now 96 mobile phone contracts for every 100 people on earth, making mobile interventions a highly viable method for extending care beyond traditional methods. Text messaging or short message service (SMS) is the most widely available mode of mobile communication and despite its simplicity, has been proven to be a reliable and effective method to induce behavior change across behavioral health targets, including problem drinking. However, large scale randomized controlled trials are needed to provide the necessary empirical evidence to validate SMS interventions and understand the mediators and moderators of outcome for help seeking heavy drinkers who are using or unable to attend in-person care.

DETAILED DESCRIPTION:
The study entitled, Tailored Adaptive Mobile Messaging to Reduce Problem Drinking (PD) is designed to develop and test a tailored adaptive text messaging/short message service (SMS) intervention for individuals interested in reducing their alcohol consumption.

According to the National Institute on Alcohol Abuse and Alcoholism, problem or risky drinking is defined as greater than 7 standard drinks per week for women and 14 standard drinks per week for men. Other groups have other criteria (e.g., 10 drinks for women and 14 for men per week). The Institute of Medicine reports that problem drinkers are those with mild-to-moderate problem severity who do not have physical dependence.

Heavy drinking individuals with non-abstinence goals rarely seek treatment for excessive alcohol use, and newer methods such as internet screening and mobile apps provide opportunities to engage and treat this difficult to reach population. There are now 96 mobile phone contracts for every 100 people on earth, making mobile interventions a highly viable method for extending care beyond traditional methods. Text messaging or short message service (SMS) is the most widely available mode of mobile communication and despite its simplicity, has been proven to be a reliable and effective method to induce behavior change across behavioral health targets, including problem drinking. However, large scale randomized controlled trials are needed to provide the necessary empirical evidence to validate SMS interventions and understand the mediators and moderators of outcome for help seeking heavy drinkers who are using or unable to attend in-person care.

The investigators recently completed an R34 study to develop the first automated tailored adaptive (TA) text messaging intervention for problem drinking (PD) adults (Muench et al. 2017). The study compared TA to different automated once a day static messaging including: tailored only messaging (TO), loss framed messaging (LF), gain frame messaging (GF), and weekly mobile assessment only (MA) over 12 weeks in 171 problem drinkers recruited on the internet across the US. All messaging groups outperformed MA on most drinking outcomes, and the TA group had the largest effect sizes on every drinking outcome, with an average weekly drink reduction of 9 standard drinks at week 12. Over an 8-month period, 1149 individuals across the country took the web-based screening survey, highlighting the demand for messaging in this population. Furthermore, 94.7% of participants (Ps) enrolled completed the end of messaging week 12 survey and 80% wanted to continue messaging following the pilot trial. There were no adverse events in this study.

Primary hypotheses:

1. The TA group will have significantly reduced weekly sum of standard drinks (SSD) and heavy drinking days (HDD) compared to MA at all time periods.
2. TO will have significantly reduced SSD and HDD compared to MA at all time points.
3. TA group will have significantly reduced SSD compared to TO at all time periods except one month follow-up.
4. Severity will moderate the relationship between TA, MA and TO and drinking in that high severity P's will make significantly greater changes in the TA group.

Exploratory aims include testing other outcomes such as drinking related consequences by group, moderators such as gender and ethnicity, and mediators such as intervention relevance and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. be fluent and able to read in English at the eighth grade level;
2. be between the ages of 21 and 75;
3. have an estimated average weekly consumption of greater than 9 or 11 standard drinks per week for women and men, respectively OR at least two nights a week of drinking more than 4 drinks in one sitting for women and 5 drinks for men.
4. be willing to reduce their drinking to non-hazardous levels;
5. be willing to provide informed consent;
6. own a mobile phone, have an active email address, are willing to receive and respond to up to 115 text messages total per month (average = 50); and
7. give the name of a collateral who can be contacted in case of loss of contact or emergency.

Exclusion Criteria:

1. present with significant substance use or a current substance use disorder (for any substance other than alcohol, nicotine, or caffeine), which is defined as greater than once weekly use in the past month/more than twice weekly use of marijuana;
2. present with a serious psychiatric illness or suicide risk as measured by previous inpatient treatment, medications for psychosis or recent suicidality;
3. demonstrate clinically severe alcoholism, as evidenced by physical withdrawal symptoms or a history of serious withdrawal symptoms (e.g., hallucinations, seizures, or delirium tremens), and score greater than 12 on the Short Alcohol Withdrawal Scale (SAWS).
4. report a medical condition that precludes drinking any alcohol; or
5. demonstrate cognitive impairment as evidenced by a score of less than 7 out of 10 on the consent form quiz.
6. express a desire to abstain or intent to obtain additional substance abuse treatment while in the study;

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Standard drinks | 6 months
  Weekly sum of standard drinks (SSD)
Heavy days | 6 months
  Heavy drinking days (HDD)

SECONDARY OUTCOMES:
Weekly drinking | 6 months
  Drinking days per week
Daily drinking | 6 months
  Drinks per drinking day
Consequences | 6 months
  Drinking related consequences

CONTACTS AND LOCATIONS:
Locations (1):
- Partnership for Drug-Free Kids, New York, New York, United States